CLINICAL TRIAL: NCT06960447
Title: Comparative Efficacy of Nd:YAG and Alexandrite Laser Treatments in Hidradenitis Suppurativa: A Split-Person, Non-Inferiority Study
Brief Title: Nd:YAG vs Alexandrite Laser Treatment in Hidradenitis Suppurativa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Mickey Horissian, Assistant Professor of Dermatology, Geisinger Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0947
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-05

CONDITIONS: Hidradenitis Suppurativa (HS)
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: Split-person trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Receiving treatment with both laser types (Experimental): Participants will receive split-body treatment, receiving Nd:YAG laser treatment to an affected anatomical site (axilla, inframammary region, or groin) and Alexandrite laser to the contralateral side. The treatment side will be randomized and maintained through the study.
  Interventions: Device: Nd:YAG Laser; Device: Alexandrite Laser

INTERVENTIONS:
Device: Nd:YAG Laser — Nd:YAG laser applied to one side of the participant's body (e.g. left or right) according to randomization, every 4-6 weeks for 4 consecutive treatments.
Device: Alexandrite Laser — Alexandrite laser applied to the contralateral side of the participant's body (e.g. left or right) according to randomization, every 4-6 weeks for 4 consecutive treatments.

SUMMARY:
The purpose of this study is to evaluate whether Alexandrite laser treatment is non-inferior to Nd:YAG (neodymium-doped yttrium aluminum garnet) laser treatment of hidradenitis suppurativa (HS).

ELIGIBILITY:
Inclusion Criteria:

* Geisinger male or female patients with a diagnosis of hidradenitis suppurativa (all stages of disease)
* 12-75 years of age
* Not on concurrent systemic therapy (e.g., antibiotics, biologic therapies)
* Must have not used systemic therapies within 2 weeks of enrollment in study
* Able and willing to provide consent

Exclusion Criteria:

* Patients who cannot tolerate laser therapy
* Patients who cannot wear protective eyewear
* Patients who are pregnant

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
HiSCR50 | 6 months
  Percentage of patients achieving a 50% reduction in their hidradenitis suppurativa clinical response (HiSCR) score.
HiSQOL | 6 months
  The Hidradenitis Suppurativa Quality Of Life (HiSQOL) scale, a validated HS quality of life index and is comprised of a 17-item HS-specific HRQOL instrument with a 7-day recall period. Score ranges from 0 to 68, with higher scores indicating more severe impact

SECONDARY OUTCOMES:
Pain VAS score | 6 months
  Visual analogue score for pain ranging from 0-10 with higher scores indicating worse pain.
Pruritus numeric rating scale | 6 months
  As measured by a numeric rating scale from 0-10 with higher scores indicating worse itching.
Days free of disease in last 30 days | 6 months
  The number of days a patient has not had a flare of HS in the past 30 days.
AN Count | 6 months
  Number of abscesses and nodules on exam

CONTACTS AND LOCATIONS:
Overall Officials: Mikael K Horissian, MD, Principal Investigator — Geisinger Clinic

IPD SHARING:
Plan to Share IPD: No